CLINICAL TRIAL: NCT05285033
Title: Real-world Effectiveness and Treatment Sequences in Patients With Extensive Stage SCLC Who Received Lurbinectedin as Part of the French Early Access Program (ATU).
Brief Title: RW Effectiveness of Lurbinectedin in Extensive Stage SCLC
Acronym: LURBICLIN
Status: Completed | Type: Observational
Sponsor: Intergroupe Francophone de Cancerologie Thoracique (Other)
Collaborators: Groupe Francais De Pneumo-Cancerologie (Other); PharmaMar (Industry)
Responsible Party: Sponsor
Other Study IDs: IFCT-2105
Record Dates: First submitted 2022-03-04; First posted 2022-03-17 (Actual); Last update posted 2023-01-06 (Actual); Status verified 2023-01

CONDITIONS: Small-cell Lung Cancer
Keywords: IFCT; Small-cell Lung Cancer; Lurbinectedin; Real-world study
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — PM 01183

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Lurbinectedin — Patients who received at least one dose of treatment with lurbinectedin as part of the French Early Access Program (ATU program).

SUMMARY:
LURBICLIN cohort will describe the demographic and clinical characteristics of patients who received at least one dose of lurbinectedin as part of ATU program. LURBICLIN will evaluate effectiveness and safety of lurbinectedin in real-world conditions.

DETAILED DESCRIPTION:
LURBICLIN cohort will describe the demographic and clinical characteristics of patients who received at least one dose of lurbinectedin as part of ATU program. LURBICLIN will evaluate overall survival, real world progression-free survival, best response and duration of treatment in patients with advanced, metastatic Small Cell Lung Cancer (SCLC) who received lurbinectedin as part of the French Early Access Program (ATU). Previous and subsequent treatments (treatment delivered immediately after treatment with lurbinectedin) will be recorded. Those outcomes will be correlated to clinical, pathological, and radiological characteristics of patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically or cytologically confirmed extensive stage Small Cell Lung Cancer
* Patients who were informed about the study and accepted for their data to be collected
* Patients who received at least one dose of treatment with lurbinectedin as part of the French Early Access Program (ATU program).
* Selection period spans from June 2020 until March 2021 for initiation of treatment with lurbinectedin.

Exclusion Criteria:

* Patients enrolled in a clinical trial assessing treatment with lurbinectedin

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with histologically or cytologically confirmed extensive stage Small Cell Lung Cancer who received at least one dose of treatment with lurbinectedin as part of the French Early Access Program (ATU program).
Sampling Method: Non-Probability Sample
Enrollment: 312 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-12-15 (Actual); Study Completion 2022-12-15 (Actual)

PRIMARY OUTCOMES:
demographic and clinical characteristics of patients | 8 months
  age
demographic and clinical characteristics of patients | 8 months
  sex
demographic and clinical characteristics of patients | 8 months
  clinical stage
demographic and clinical characteristics of patients | 8 months
  prior therapy

SECONDARY OUTCOMES:
Overall Survival (OS) | 8 months
  OS is defined as the time from the first dose of treatment with lurbinectedin to death from any cause
Real-world progression-free survival | 8 months
  time from first dose of treatment with lurbinectedin to first occurrence of disease progression or death from any cause during the study
Best response | 8 months
  best response recorded from the start of treatment with lurbinectedin until disease progression or start of further anti-cancer treatment
Duration of treatment | 8 months
  time from first dose of treatment to discontinuation of treatment (interruption of more than 2 months) with lurbinectedin
Pattern of tumor progression | 8 months
  site of disease progression after treatment with lurbinectedin
Duration of treatment with lurbinectedin beyond progression | 8 months
  time between first occurrence of disease progression and treatment discontinuation
Adverse Drug Reaction | 8 months
  maximal grade 3-4-5 treatment-related adverse events (SAEs, TRAEs), and immune-related events will be recorded for each patient

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Girard, Study Chair — Institut Curie
Locations (2):
- France (2):
  - Institut Curie, Paris
  - Villefranche-Sur-Saône - CH, Villefranche-sur-Saône

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Trigo J, Subbiah V, Besse B, Moreno V, Lopez R, Sala MA, Peters S, Ponce S, Fernandez C, Alfaro V, Gomez J, Kahatt C, Zeaiter A, Zaman K, Boni V, Arrondeau J, Martinez M, Delord JP, Awada A, Kristeleit R, Olmedo ME, Wannesson L, Valdivia J, Rubio MJ, Anton A, Sarantopoulos J, Chawla SP, Mosquera-Martinez J, D'Arcangelo M, Santoro A, Villalobos VM, Sands J, Paz-Ares L. Lurbinectedin as second-line treatment for patients with small-cell lung cancer: a single-arm, open-label, phase 2 basket trial. Lancet Oncol. 2020 May;21(5):645-654. doi: 10.1016/S1470-2045(20)30068-1. Epub 2020 Mar 27. PMID 32224306
- See also: IFCT website — https://www.ifct.fr/etudes-cliniques/806-ifct-2105